CLINICAL TRIAL: NCT00659854
Title: Cow's Milk Allergy in Infants With Obstructive Sleep Apnea
Brief Title: Cow's Milk Allergy in Infants With Obstructive Sleep Apnea (OSA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Aviv D Goldbart MD, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOR467908CTIL
Record Dates: First submitted 2008-04-07; First posted 2008-04-16 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-04

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: obstructive sleep apnea syndrome; The study examines the response of infants diagnosed with obstructive sleep apnea syndrome to diet changes
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non milk or soy based formula (Placebo Comparator): 25 infants , non milk or soy based formula .
  Interventions: Dietary Supplement: Non milk or soy based formula
- 2 (Active Comparator): Intervention with milk based formula will be given to 25 infants.
  Interventions: Dietary Supplement: milk based formula

INTERVENTIONS:
Dietary Supplement: Non milk or soy based formula — Babies will be given a non milk or soy base formula for 12 weeks
  Arms: Non milk or soy based formula
Dietary Supplement: milk based formula — Babies will be given a milk based formula for 12 weeks
  Arms: 2

SUMMARY:
Cow's milk allergy may be involved in the evolution of sleep apnea in infants. The study will assess the effects of specifies diet changes (i.e. non-milk based formula) on the infant. Specifically , infants will be investigated by sleep studies in order to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Polysomnographically diagnosed OSA
2. Age is 2-24 months
3. Clinical suspicion of milk allergy due to findings in the medical history or physical exam

Exclusion Criteria:

1. Congenital defects in the pulmonary and gastrointestinal systems
2. Family history of genetic diseases or familial syndromes
3. Infantile asthma.

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Polysomnographic variables following 12 weeks of non-milk based formula, in comparison to baseline(prior to diet change). | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Aviv D Goldbart, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka University Medical center, Beersheba, Israel